CLINICAL TRIAL: NCT06162793
Title: eHealth for Promoting Regular Physical Activity in Medical Rehabilitation Maintenance: the RehaPlus+ Concept
Brief Title: eHealth for Promoting Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eHealth_RehaPlus_01
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: rehabilitation; eHealth; mHealth; telemedicine; cardiovascular disease
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RehaPlus+ (Experimental): Customized motivational text messages twice weekly for six months
  Interventions: Behavioral: RehaPlus+
- Usual care (No Intervention): Standard care (Six-month German outpatient program "IRENA")

INTERVENTIONS:
Behavioral: RehaPlus+ — 24-week eHealth intervention
  Arms: RehaPlus+

SUMMARY:
Coronary artery disease (CAD) is a chronic disease without a definitive cure. Cardiac rehabilitation (CR) is a class IA recommendation for CAD patients, that focuses on risk factor reduction and physical exercise. It comprises three stages: Phase I in the acute setting, Phase II for reconditioning, and Phase III as maintenance. Despite the effectiveness of Phase II, there is often a decline in cardiovascular risk profiles afterward due to lifestyle challenges and inadequate support.

Traditional maintenance programs face limitations, such as high costs and patient-related barriers. With the increasing prevalence of mobile devices and digitalization, eHealth can enhance rehabilitation effectiveness post-discharge. Previous studies support the effectiveness of eHealth in CR maintenance.This study aims to evaluate the effectiveness of the eHealth program "RehaPlus+" in motivating CAD patients for increased physical activity (PA).

DETAILED DESCRIPTION:
Coronary artery disease (CAD), a chronic disease lacking a definitive cure, can be mitigated through cardiac rehabilitation (CR). As a class IA recommendation for CAD patients, CR employs evidence-based therapy to minimize the physiological and psychological impacts of CAD, reduce morbidity and mortality rates, and enhance physical performance. CR involves three stages: Phase I for acute intervention, Phase II for reconditioning, and Phase III for maintenance. Despite the effectiveness of Phase II CR, cardiovascular risk profiles often deteriorate thereafter, attributed to the challenge of maintaining a healthy lifestyle and limited support of patients. Traditional maintenance programs face barriers such as high costs and time constraints while the COVID-19 pandemic further disrupted on-site programs.The rise of eHealth solutions, such as the RehaPlus+ concept, driven by innovative technologies and the prevalence of mobile devices, aligns with the trend of digitalization in healthcare. This evolution presents opportunities to enhance patient health maintenance, with eHealth applications amplifying rehabilitation effectiveness post-discharge. Previous studies support the efficacy of eHealth in CR maintenance.

This study aims to assess the effectiveness of the eHealth program "RehaPlus+" in supporting CAD patients for increased physical activity (PA). The hypothesis is that RehaPlus+ will be as effective as the German standard center-based program ("IRENA") in supporting regular PA, Activity of Daily Living (AoDL), and improving psychological well-being, cardiac self-efficacy (CSE), health-related well-being, and work ability six months after Phase II CR discharge.

The study will include patients with CAD allocated to either a 24-week eHealth group (RehaPlus+) or a conventional outpatient program group (IRENA) using a quasi-experimental approach. RehaPlus+ recipients will receive customized motivational text messages twice weekly for six months, while the IRENA group will engage in a six-month outpatient program involving 24 sessions of 90-minute strength and endurance training. The primary outcomes, evaluated using the BSA questionnaire, will focus on regular PA and weekly activities of daily living (AoDL) six months post-rehabilitation. Secondary outcomes will examine physical activity during work and floors climbed weekly (BSA), psychological well-being (WHO-5), cardiac self-efficacy (CSE), health-related well-being (SF-36), and work ability (WAI) via questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* documented coronary artery disease
* referral to inpatient rehabilitation
* signed informed consent

Exclusion Criteria:

* language barriers
* incapable of understanding study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Physical Activity | week 24
  Physical activity will be assessed by the German "Physical Activity and Sports questionnaire" (BSA). The minimum value is 0, the maximum value is unlimited. A higher value indicates a better outcome.
Activity of Daily Living | week 24
  Activity of Daily Living will be assessed by the German "Physical Activity and Sports questionnaire" (BSA). The minimum value is 0, the maximum value is unlimited. A higher value indicates a better outcome.

SECONDARY OUTCOMES:
Change in Work requirements and workload | Baseline and week 24
  Work requirements and workload will be assessed using the "Workability Index (WAI)" questionnaire. The minimum value is 7, and the maximum value is 49, where a higher value indicates improved work ability.
Change in Health-related quality of life | Baseline and week 24
  Health-related quality of life will be assessed using the SF-36 questionnaire. The minimum value is 0, and the maximum value is 100, where a higher value signifies greater well-being.
Change in Wellbeing | Baseline and week 24
  Wellbeing will be assessed using the "WHO-5 Well-Being Index". The minimum value is 0, and the maximum value is 25, where a higher value signifies greater well-being.
Change in Cardiac Self-Efficacy (CSE) | Baseline and week 24
  Cardiac self-efficacy will be measured using the Cardiac Self-Efficacy questionnaire. The minimum value is 0, and the maximum value is 100, where a higher value signifies greater well-being.
Physical activity (PA) at work | week 24
  Physical activity at work will be assessed by the German "Physical Activity and Sports questionnaire" (BSA). The minimum value is 0, the maximum value is 9. A higher value indicates a better outcome.
Climbed floors | week 24
  Climbed floors will be assessed by the German "Physical Activity and Sports questionnaire" (BSA). The minimum value is 0, the maximum value is unlimited. A higher value indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Königsfeld, Ennepetal, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Heimer M, Schmitz S, Teschler M, Schafer H, Douma ER, Habibovic M, Kop WJ, Meyer T, Mooren FC, Schmitz B. eHealth for maintenance cardiovascular rehabilitation: a systematic review and meta-analysis. Eur J Prev Cardiol. 2023 Oct 26;30(15):1634-1651. doi: 10.1093/eurjpc/zwad145. PMID 37154363
- [Derived] Waranski M, Garbsch R, Kotewitsch M, Teschler M, Schmitz B, Mooren FC. A Behavioral Change-Based Mobile Intervention for Promoting Regular Physical Activity in Medical Rehabilitation Maintenance of Patients With Coronary Artery Disease: Controlled Trial. J Med Internet Res. 2024 Oct 8;26:e56480. doi: 10.2196/56480. PMID 39378432